CLINICAL TRIAL: NCT05515796
Title: Clinical Application of Efficacy Prediction Model Based on Epigenetics Multi-omics Sequencing in Neoadjuvant Immunotherapy of Gastrointestinal Tumors
Brief Title: Multi-omics Sequencing in Neoadjuvant Immunotherapy of Gastrointestinal Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, wang bin, Director of Gastroenterology, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DP-GE-ICI
Record Dates: First submitted 2022-08-20; First posted 2022-08-25 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Immunotherapy; Gastric Cancer; Rectal Cancer; Chemotherapy Effect; Radiotherapy
Keywords: Immunotherapy; Gastric Cancer; Rectal Cancer; neoadjuvant; Terelizumab (aka Tislelizumab); radiotherapy; oxaliplatin; capecitabine
MeSH Terms: conditions — Stomach Neoplasms; Rectal Neoplasms | interventions — Trastuzumab; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Gastric cancer:CapeOx+Terelizumab (aka Tislelizumab)(HER2 negative)（n=80） Gastric cancer:CapeOx+Trastuzumab+Terelizumab (aka Tislelizumab) (HER2 positive )（n=20） Rectal cancer:Radiotherapy with CapeOx+ Terelizumab (aka Tislelizumab)（n=100）
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Gastric cancer:CapeOx+Terelizumab (aka Tislelizumab)(HER2 negative) (Experimental): CapeOx+Terelizumab (aka Tislelizumab)(HER2 negative):
  Cycle 1 up to Cycle 3 CapeOX + Terelizumab (aka Tislelizumab) therapy Cycle: Day 1 through Day 21
  Interventions: Drug: Terelizumab (aka Tislelizumab); Drug: CapeOx
- Gastric cancer:CapeOx+Trastuzumab+Terelizumab (aka Tislelizumab) (HER2 positive ) (Experimental): CapeOx+Trastuzumab+Terelizumab (aka Tislelizumab) (HER2 positive ):
  Cycle 1 up to Cycle 3 CapeOx+Trastuzumab+Terelizumab (aka Tislelizumab) Cycle: Day 1 through Day 21
  Interventions: Drug: Terelizumab (aka Tislelizumab); Drug: CapeOx; Drug: Trastuzumab
- Rectal cancer:Radiotherapy with CapeOx+ Terelizumab (aka Tislelizumab) (Experimental): Rectal cancer:
  Cycle 1:25 Gy/5 fractions (Day 1 through Day 7) Cycle 2 up to Cycle 3 CapeOX + Terelizumab (aka Tislelizumab) therapy(Day 1 through Day 21)
  Interventions: Drug: Terelizumab (aka Tislelizumab); Drug: CapeOx; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Terelizumab (aka Tislelizumab) — q3w Terelizumab (aka Tislelizumab) 200mg on day 1 of each cycle
Drug: CapeOx — Oxaliplatin(130mg/m2) on day 1 of each cycle and Capecitabine:Dose of 1000mg/m2,14days
Drug: Trastuzumab — q3w Trastuzumab (6 mg/kg following an initial loading dose of 8 mg/kg) on day 1 of each cycle
  Arms: Gastric cancer:CapeOx+Trastuzumab+Terelizumab (aka Tislelizumab) (HER2 positive )
Radiation: Radiotherapy — 25 Gy/5 fractions
  Arms: Rectal cancer:Radiotherapy with CapeOx+ Terelizumab (aka Tislelizumab)

SUMMARY:
immunotherapy，gastric cancer，rectal cancer，biomark

DETAILED DESCRIPTION:
To investigate the effect of Terelizumab (aka Tislelizumab) combined with XELOX in Neoadjuvant Therapy for gastrointestinal tumors.

To explore new biomarkers that can predict the efficacy of combined immunotherapy, and to establish a clinical efficacy prediction model by means of bioinformatics to prospectively judge the efficacy and guide the follow-up individualized and accurate treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patients are able to understand and voluntarily sign the written informed consent, which must be signed prior to the implementation of the designated research procedures required by the study.
* The age at the time of signing the informed consent form (ICF) is ≥ 18 years old, both male and female.
* Locally advanced or metastatic gastric / gastroesophageal junction adenocarcinoma (clinical stage ≥ T2N0M0) and pMMR/MSS(tumor biopsy immunohistochemical identified pMMR or next generation sequencing identified MSS) locally advanced rectal adenocarcinoma (clinical stage T3-4N0M0 or T1-4N+M0 ) were diagnosed by comprehensive evaluation.
* The patients are willing to provide fresh tissue for biomarker analysis, and the tissue samples provided are of sufficient quality to evaluate the status of biomarkers. If sufficient tissue is not provided, repeated sampling may be required.
* The patient has an Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 or 1.
* The expected survival time was ≥ 3 months.
* The patient has adequate organs function

  1. The patient has adequate hematologic function, as evidenced by an absolute neutrophil count (ANC) ≥1.5*10^9/L, hemoglobin ≥90g/L (5.58 mmol/L), and platelets ≥100*10^9/L.
  2. The patient has adequate renal function as defined by a serum creatinine ≤1.5 times the ULN, or creatinine clearance (measured via 24-hour urine collection) ≥50 mL/minute (that is, if serum creatinine is >1.5 times the ULN, a 24-hour urine collection to calculate creatinine clearance must be performed).
  3. The patient has adequate hepatic function as defined by a total bilirubin ≤1.5 mg/dL (25.65 μmol/L), and aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 times the upper limit of normal (ULN; or 5.0 times the ULN in the setting of liver metastases).
  4. The patient must have adequate coagulation function as defined by international normalized ratio (INR) ≤1.5
* Within 7 days before the first administration, women of childbearing age must confirm that the serum pregnancy test is negative and agree to use effective contraceptives during the study period and within 180 days after the last administration. In this program, women of childbearing age are defined as sexually mature women:

  1. No hysterectomy or bilateral ovariectomy
  2. Natural menopause does not last for 24 months (amenorrhea after cancer treatment does not rule out fertility) (that is, menstruation occurs at any time in the previous 24 months).

For male patients whose sexual partners are women of childbearing age, they must agree to use effective contraception during the study drug use and within 180 days after the last administration.

Exclusion Criteria:

* Palliative local treatment was given to non-target lesions within 2 weeks before the first administration, and systemic non-specific immunomodulatory therapy (such as interleukin, interferon, thymosin, etc.) was received within 2 weeks before the first administration. Chinese herbal medicine or proprietary Chinese medicine with anti-tumor indications was received within 2 weeks before the first administration.
* The patient has previously received immune checkpoint inhibitors (such as anti-PD-1 antibodies, anti-PD-L1 antibodies, anti-CTLA-4 antibodies, etc.), immune checkpoint agonists (such as antibodies against ICOS, CD40, CD137, GITR, OX40 targets, etc.), immune cell therapy, etc. any treatment aimed at the immune mechanism of tumor.
* There was a history of gastrointestinal perforation and gastrointestinal fistula within 6 months before the first administration. If the perforation or fistula has been removed or repaired, and the disease has been judged by the researchers to recover or remission, it may be allowed to join the group.
* Active or previously recorded inflammatory bowel disease (such as Crohn's disease or ulcerative colitis). Unable to swallow, malabsorption syndrome, or uncontrollable nausea, vomiting, diarrhea or other gastrointestinal diseases that seriously affect drug use and absorption.
* There were active malignant tumors in the past 3 years, except for tumors that participated in the study and local tumors that had been cured. such as skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ, breast cancer in situ, localized prostate cancer and so on.
* Active or untreated brain metastases, meningeal metastases, spinal cord compression or leptomeningeal diseases are known.

However, the patients who met the following requirements and had measurable lesions outside the central nervous system were allowed to enter the group: asymptomatic after treatment, imaging was stable for at least 4 weeks before the start of treatment (such as no new or enlarged brain metastases). And systemic corticosteroids and anticonvulsant drugs have been stopped for at least 2 weeks.

* There are pleural effusion with clinical symptoms, pericardial effusion or ascites requiring frequent drainage (≥ 1 / month).
* Study active autoimmune diseases that require systematic treatment within 2 years before the start of treatment, or researchers determine the existence of autoimmune diseases that may recur or plan treatment. Except for the following:

  1. Skin diseases that do not require systematic treatment (e.g. vitiligo, hair loss, psoriasis or eczema)
  2. Hypothyroidism caused by autoimmune thyroiditis requires only a stable dose of hormone replacement therapy.
  3. Type I diabetes mellitus requiring only a stable dose of insulin replacement therapy
  4. Asthma has been completely relieved in childhood and no intervention is needed in adults.
  5. The researchers determined that the disease would not recur without external triggers.
* There are any of the following cardio-cerebrovascular diseases or cardio-cerebrovascular risk factors:

  1. Within 6 months before the first administration, there were myocardial infarction, unstable angina pectoris, cerebrovascular accident, transient ischemic attack, acute or persistent myocardial ischemia, symptomatic heart failure (according to New York Heart Association functional grade 2 or above), symptomatic or poorly controlled arrhythmia, or any arterial thromboembolic event.
  2. There was a history of deep venous thrombosis, pulmonary embolism or other severe thromboembolism within 3 months before the first administration.
  3. There are major vascular diseases, such as aortic aneurysm, aortic dissecting aneurysm, internal carotid artery stenosis, which may be life-threatening or require surgery within 6 months.
  4. Previous history of myocarditis and cardiomyopathy.
  5. Left ventricular ejection fraction (LVEF) < 50%.
* Toxicity that has not been alleviated by previous antineoplastic therapy is defined as undiminished to Grade 0 or 1 of the National Cancer Institute (NCI) General terminology Standard for adverse events (CTCAE) (NCICTCAEv5.0), or to the level specified in the selection / exclusion criteria, with the exception of alopecia / pigmentation. The patients who develop irreversible toxicity and are not expected to increase after drug administration (such as hearing loss) may be included in the study after consultation with researchers. Long-term toxicity caused by radiotherapy may be included in the study after consultation with the researchers who are determined by the researchers to be unable to recover.
* Grade 2 peripheral nerve disease was defined according to NCI CTCAE v5.0 standard.
* Interstitial lung disease or non-infectious pneumonia is known to be symptomatic or requires systemic glucocorticoid treatment in the past, and researchers have determined that it may affect toxicity assessment or management associated with research treatment.
* Active tuberculosis is known to exist. The patients suspected of having active pulmonary tuberculosis should be examined for chest X-ray, sputum and excluded by clinical symptoms and signs.
* Received systemic anti-infective therapy (excluding antiviral therapy for hepatitis B or C) within 2 weeks before the first administration.
* The history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation are known.
* There are clinical active hemoptysis, active diverticulitis, abdominal abscess and gastrointestinal obstruction.
* There were significant clinical bleeding symptoms or definite bleeding tendency within 1 month before the first administration, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, or vasculitis.
* It is known that endoscopy shows signs of active bleeding.
* There were other major operations in addition to the diagnosis of gastric cancer within 28 days before the first administration.
* Untreated active hepatitis B patients (HBsAg positive and HBV-DNA more than 1000 copies / ml [200IU/ml] or higher than the detection lower limit), patients with hepatitis B were required to receive anti-HBV treatment during the study treatment; active hepatitis C patients (HCV antibody positive and HCV-RNA levels higher than the detection lower limit).
* Those who are known to have a history of immunodeficiency or are HIV positive.
* Known active syphilis infection.
* Is participating in another clinical study, unless it is a follow-up period for observational, non-interventional clinical studies or interventional studies.
* The patients who needed systemic treatment with glucocorticoids (> 10mg/ prednisone or equivalent dose) or other immunosuppressive drugs within 14 days before the first administration. Except for the following:

  1. If there is no active autoimmune disease, inhaled, ophthalmic or topical glucocorticoids or doses of ≤ 10mg/ prednisone or equivalent doses of other glucocorticoids are allowed.
  2. Physiological dose of systemic glucocorticoid ≤ 10mg/ prednisone or equivalent dose of other glucocorticoids.
  3. Glucocorticoids are used as pretreatment of infusion-related reactions or allergic reactions (such as medication before CT examination).
* The live vaccine was given within 30 days of the first administration, or is planned during the study period.
* A history of severe hypersensitivity to other monoclonal antibodies is known.
* It is known to be unable to meet the requirements of the trial because of mental illness or substance abuse disorder.
* The patients who are known to have a history of allergy or hypersensitivity to drugs or any of its components in the combined immunotherapy regimen.
* The patient is pregnant or breastfeeding.
* The researchers believe that there may be a risk of receiving the study drug treatment, or any condition that will interfere with the evaluation of the study drug or the safety of the patients or the interpretation of the research results.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | 6 months
  Pathological complete response will be evaluated with American Joint Committee on Cancer (AJCC) Cancer Staging

SECONDARY OUTCOMES:
Major pathologic response (MPR) | 6 months
  It is defined as residual tumors less than 10% after neoadjuvant immunotherapy and(or) chemotherapy
Overall survival (OS) | 2 years
  Time from study entry to death from any cause.
Disease-free survival (DFS) | 2 years
  Time from study entry to disease recurrence or patient death due to disease progression
R0 resection rate | 6 months
  Rate of microscopically margin-negative resection

OTHER OUTCOMES:
Correlation analysis of evaluating the relationship between clinicopathological characteristics and neoadjuvant immunochemotherapy efficacy | 2 years
  Correlation analysis of evaluating the relationship between clinicopathological characteristics and neoadjuvant immunochemotherapy efficacy
Correlation analysis of evaluating the relationship between multi-omics analysis of tumor tissue and neoadjuvant immunochemotherapy efficacy | 2 years
  Correlation analysis of evaluating the relationship between multi-omics analysis of tumor tissue and neoadjuvant immunochemotherapy efficacy
EORTC QLQ-C30(V3) | 2 years
  Gastric cancer and rectal cancer：The EORTC Core Quality of Life questionnaire (EORTC QLQ-C30) is designed to measure cancer patients' physical, psychological and social functions.
EORTC QLQ-STO22 | 2 years
  EORTC Quality of Life Questionnaire - Gastric Cancer Module:to be used in conjunction with the EORTC QLQ-C30 to assess health-related quality of life in gastric cancer.
EORTC QLQ-CR29 | 2 years
  EORTC Quality of Life Questionnaire - Colorectal Cancer Module:to be used in conjunction with the EORTC QLQ-C30 to assess quality of life in patients with colorectal cancer

CONTACTS AND LOCATIONS:
Overall Officials: wang bin, Principal Investigator — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Locations (1):
- Army Medical Center, Chongqing, Other (Non U.s.), China

IPD SHARING:
Plan to Share IPD: Undecided